



| NCT Number: NCT05252702 |
|-------------------------------------------|
| Aveir <sup>™</sup> DR i2i Study |
| Aveir Dual-Chamber Leadless i2i IDE Study |
| Study Document No: ABT-CIP-10416 |
| Version C |
| Date: 12-AUG-2022 |

Sponsor Abbott Medical

Cardiac Rhythm Management 15900 Valley View Court Sylmar, CA 91342

Template Page 1 of 1

## **Statistical Analysis Plan**

# ABT-CIP-10416/ Ver C CRD 1023

Aveir<sup>TM</sup> DR i2i Study

Aveir Dual Chamber Leadless i2i study

## **Statistical Analysis Plan (SAP)**

Version C

August 12, 2022

Template 



## **Statistical Analysis Plan**

## **TABLE OF CONTENTS**

| SYNOPSIS OF STUDY DESIGN4 | | |
|---|---|---|
| Purpose of the Statistical Analysis Plan | | |
| Clinical Investigation Objectives | | |
| Clir | nical Investigation Design | 4 |
| End | dpoints | 4 |
| .4.1 | Primary Safety Endpoint | 4 |
| .4.2 | Primary Effectiveness Endpoint #1 | 5 |
| .4.3 | Primary Effectiveness Endpoint #2 | 5 |
| .4.4 | Secondary Safety Endpoint | 5 |
| .4.5 | Secondary Effectiveness Endpoint | 5 |
| Rar | ndomization | 5 |
| Blin | ding | 5 |
| ANAL | YSIS CONSIDERATIONS | 5 |
| Ana | alysis Populations | 5 |
| .1.1 | Full Analysis Population | 5 |
| Sta | tistical Methods | 5 |
| .2.1 | Descriptive Statistics for Continuous Variables | 6 |
| .2.2 | Descriptive Statistics for Categorical Variables | 6 |
| .2.3 | Survival Analyses | 6 |
| End | lpoint Analysis | 6 |
| .3.1 | Primary Safety Endpoint Analysis | 6 |
| .3.2 | Primary Effectiveness Endpoint #1 Analysis | 7 |
| .3.3 | Primary Effectiveness Endpoint #2 Analysis | 8 |
| .3.4 | Secondary Safety Endpoint Analysis | <u>S</u> |
| .3.5 | Secondary Effectiveness Endpoint Analysis | g |
| Sar | nple Size Calculations | 11 |
| Inte | rim Analysis | 12 |
| 2.7 Study/Trial Success | | 12 |
| 2.8 Subgroups for Analysis | | 13 |
| Har | ndling of Missing Data | 13 |
| 2.10 Poolability Issue | | 14 |
| | Pur Clir Clir End. 4.1 4.2 4.3 4.4 4.5 Rar Blin ANAL Ana. 1.1 Sta 2.1 2.2 2.3 End. 3.1 3.2 3.3 5 Sar Interest Stu Substitute Substit | Purpose of the Statistical Analysis Plan Clinical Investigation Objectives Clinical Investigation Design Endpoints |



## **Statistical Analysis Plan**

| 2.12 | 2 Adjustments for Covariates | 14 |
|------|-------------------------------------------|----|
| 3.0 | DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA | 15 |
| 3.1 | Baseline and Demographic Characteristics | 15 |
| 3.2 | Adverse Events | 15 |
| 3.3 | Subject Early Termination | 15 |
| 3.4 | | |
| 3.5 | Additional Data | 15 |
| 3.6 | 24-Hour Holter Monitor Data Analysis | 16 |
| 4.0 | DOCUMENTATION AND OHER CONSIDERATIONS | 17 |
| 5.0 | ACRONYMS AND ABBREVIATIONS | 17 |
| 6.0 | REFERENCES | 17 |



## Statistical Analysis Plan

#### 1.0 SYNOPSIS OF STUDY DESIGN

#### 1.1 Purpose of the Statistical Analysis Plan

This statistical analysis plan (SAP) is intended to provide a detailed and comprehensive description of the planned methodology and analysis to be used for the ABT-CIP-10416 (CRD 1023), the Aveir DR i2i Study clinical investigation. This plan is based on the version C of the Clinical Investigation Plan (CIP).

### 1.2 Clinical Investigation Objectives

#### Primary Objectives

The primary objectives of this study are to evaluate the safety and effectiveness of the Aveir™ DR LP system through 3 months post-implant in a subject population indicated for a DDD(R) pacemaker system.

#### Secondary Objectives

The secondary objectives of this study are to evaluate the safety and effectiveness of the Aveir atrial LP through 3 months post-implant in a subject population indicated for a DDD(R) pacemaker system to support an indication for AAI(R) pacing.

#### 1.3 Clinical Investigation Design

This is a prospective, multi-center, international, single-arm, pivotal investigational study designed to evaluate the safety and effectiveness of the Aveir DR LP system in a subject population indicated for a DDD(R) pacemaker.

The clinical study will enroll up to 550 subjects from up to 85 participating centers from the United States, Canada, Europe, and Asia Pacific. The Sponsor may approach centers in other countries for participation in the clinical investigation as needed.

Subjects participating in the clinical study will be followed through at least 12 months with data collected at baseline, implant procedure, prior to hospital discharge, and follow-up at 1 month, 3 months, 6 months, 12 months and every 6 months thereafter until study completion.

## 1.4 Endpoints

The DR Study will have the following endpoints.

#### 1.4.1 Primary Safety Endpoint

The primary safety endpoint evaluates the 3-month Aveir DR LP system complication free rate (CFR) in de novo subjects based on Clinical Event Committee (CEC) adjudication of adverse events.

Template 



## **Statistical Analysis Plan**

#### 1.4.2 Primary Effectiveness Endpoint #1

The primary effectiveness endpoint #1 evaluates the 3-month composite success rate evaluating acceptable atrial pacing thresholds and P-wave amplitudes in de novo subjects.

#### 1.4.3 Primary Effectiveness Endpoint #2

The primary effectiveness endpoint #2 evaluates the 3-month AV synchrony success rate at rest while seated in de novo subjects.

### 1.4.4 Secondary Safety Endpoint

The secondary safety endpoint evaluates the 3-month Aveir atrial LP CFR in de novo subjects based on CEC adjudication of adverse events.

#### 1.4.5 Secondary Effectiveness Endpoint

The secondary effectiveness endpoint evaluates the appropriate and proportional rate response of the atrial LP in de novo subjects during graded exercise testing (CAEP protocol).

#### 1.5 Randomization

Not Applicable.

#### 1.6 Blinding

Not Applicable.

#### 2.0 ANALYSIS CONSIDERATIONS

#### 2.1 Analysis Populations

The following analysis populations are defined for the study.

#### 2.1.1 Full Analysis Population

Full Analysis population includes all subjects who have an attempted implant. An implant is considered attempted when the Aveir Introducer Sheath or Aveir dilator is inserted through the skin of the access site.

#### 2.2 Statistical Methods

For the primary and secondary endpoints, hypothesis tests will be performed. In addition, a set of additional data will be summarized by descriptive statistics or Kaplan-Meier estimates according to the type of the data.

emplate 



## **Statistical Analysis Plan**

#### 2.2.1 Descriptive Statistics for Continuous Variables

For continuous variables (e.g., age, etc.), results will be summarized with the numbers of observations, means, and standard deviations, with quartiles, minimums, maximums, and 95% confidence intervals for the means as per the table mockups.

#### 2.2.2 Descriptive Statistics for Categorical Variables

For categorical variables (e.g., gender, cardiac disease history, etc.), will be summarized with subject counts and percentages/rates, and where specified in the table mockups, with exact 95% Clopper-Pearson confidence intervals.

#### 2.2.3 Survival Analyses

For time-to-event variables, Kaplan-Meier analysis will be conducted. Subjects without events will be censored at their last known event-free time point, and for subjects with events the time to the first event will be used for the analysis. Survival estimates of the data and associated 95% confidence interval will be presented using cumulative survival and its estimated standard error (Greenwood's formula).

### 2.3 Endpoint Analysis

The primary and secondary endpoint analysis will be based on newly enrolled (de novo) subjects in the study who have an attempted implant. De novo subjects are defined as subjects that do not have an implanted pacemaker on the date of consent through the date of the Aveir LP implant.

#### 2.3.1 Primary Safety Endpoint Analysis

The primary safety endpoint evaluates the 3-month Aveir DR LP system CFR in de novo subjects based on CEC adjudication of adverse events.

A complication is defined as a device-or-procedure-related serious adverse event (SADE) which includes both Atrial LP and Ventricular LP complications and implant procedure-related complications.

The primary safety endpoint hypothesis is:

 $H_0$ : CFR ≤ 78% vs.  $H_1$ : CFR > 78%

where 78% is the performance goal (PG).

The CFR at 3 months will be estimated as a binomial proportion and one-sided 97.5% lower confidence bound (LCB) of CFR will be calculated using the normal approximation. The null hypothesis is rejected at the 2.5% significance level if the LCB exceeds the PG of 78%. The p-value from a one-sided Z-test for the binomial proportion will also be calculated and compared to the 0.025 significance level.

The primary analysis population for the primary safety endpoint analysis will be based on subjects in the full analysis population, and the analysis will be conducted on all subjects with data available for the evaluation. Subjects who withdraw from the study or die prior to the 3-month follow-up visit (lower window) without an event (SADE) will be excluded from this analysis. SADE events that occur through 3 months (90 days) will be included in the primary safety endpoint analysis.

emplate 



## Statistical Analysis Plan

To eliminate the possible impact of Covid-19 on the primary safety endpoint analysis, CEC adjudicated primary safety events (SADEs) that are related or possibly related to Covid-19 will be excluded. Additional analysis with these events included will also be provided.

#### 2.3.2 Primary Effectiveness Endpoint #1 Analysis

The primary effectiveness endpoint #1 evaluates the 3-month composite success rate (Rate<sub>EP</sub>) evaluating acceptable atrial pacing thresholds and P-wave amplitudes in de novo subjects.

The primary effectiveness endpoint #1 hypothesis is:

 $H_0$ : Rate<sub>EP</sub>  $\leq 82.5\%$  vs.  $H_1$ : Rate<sub>EP</sub> > 82.5%

where 82.5% is the performance goal. The Rate<sub>EP</sub> is the proportion of subjects who have met success criteria in the primary effectiveness endpoint #1. The acceptable ranges for sensing and pacing which define success criteria are shown in the table below:

| Parameter | Acceptable values |
|----------------|------------------------------------|
| Pacing voltage | Pacing threshold ≤ 3.0 V at 0.4 ms |
| P Sensitivity | P-wave amplitude ≥ 1.0 mV |

Success Criteria: A subject will be considered to have met the primary effectiveness #1 endpoint if: pacing threshold voltage  $\leq$  3.0 V at 0.4 ms at 3-month visit and sensed P-wave amplitude is  $\geq$  1.0 mV at the 3-month visit

For subjects that do not have P-wave amplitude measured due to active atrial fibrillation or atrial tachyarrhythmias or any other heart rhythm conditions or procedures which prevent sensing amplitude from being measured, success will be determined from pacing threshold only. For subjects that do not have pacing threshold measured, due to active atrial fibrillation or atrial tachyarrhythmias or any other heart rhythm conditions or procedures which prevent pacing threshold from being measured, success will be determined from P-wave amplitude only. Subjects that do not have P-wave amplitude and pacing voltage, both of which are unobtainable due to active atrial fibrillation or atrial tachyarrhythmias or any other heart rhythm conditions or procedures which prevent pacing threshold from being measured, will be excluded from analysis.

The Rate<sub>EP</sub> at 3 months will be estimated as a binomial proportion and the one-sided 97.5% LCB of the Rate<sub>EP</sub> will be calculated using the normal approximation. The null hypothesis is rejected at the 2.5% significance level if the LCB exceeds the PG of 82.5%. The p-value for the one-sided Z-test will be calculated and compared to the 2.5% significance level.

The primary analysis for the primary effectiveness endpoint #1 will be based on subjects in the full analysis population. Subjects with unsuccessful implants due to reasons other than atrial pacing/sensing (e.g., cardiac anatomy) will be excluded from the analysis. Subjects who don't meet pacing/sensing success criteria at 3-months or subjects with unsuccessful implant solely due to inadequate atrial LP pacing or sensing will be counted as failures. In addition, for subjects with missing 3-month pacing threshold or P-wave amplitude data, multiple imputation will be used to impute success or failure.

Template 



## Statistical Analysis Plan



#### 2.3.3 Primary Effectiveness Endpoint #2 Analysis

The primary effectiveness endpoint #2 evaluates the 3-month AV synchrony success rate (Rate<sub>AV</sub>) at rest while seated in de novo subjects.

AV synchrony success is defined as subjects with a paced or sensed ventricular beat within 300 ms following a paced or sensed atrial beat (i.e., a synchronous cycle) for at least 70% of evaluable cardiac cycles. An independent core laboratory will evaluate collected Holter data from sites and will determine AV synchrony success in subjects.

An evaluable cardiac cycle is defined as a cycle with:

- a) An identifiable P-wave or Atrial Paced Event (AP) with an identifiable R-wave or Ventricular Paced Event (VP) (1:1 conduction) OR
- b) An identifiable R-wave or VP and a confirmed absent (flatline) P-wave or AP.

The primary effectiveness endpoint #2 hypothesis is:

 $H_0$ : Rate<sub>AV</sub>  $\leq 83\%$  vs.  $H_1$ : Rate<sub>AV</sub> > 83%

where 83% is the performance goal. The Rate<sub>AV</sub> is the proportion of subjects who met success criteria in the primary effectiveness endpoint #2.

The Rate<sub>AV</sub> at 3 months will be estimated as a binomial proportion and one-sided 97.5% LCB of the Rate<sub>AV</sub> will be calculated using the normal approximation. The null hypothesis is rejected at the 2.5% significance level if the LCB exceeds the PG of 83%. The p-value for the one-sided Z-test will be calculated and compared to the 2.5% significance level.

The primary analysis for the primary effectiveness endpoint #2 will be based on subjects in the full analysis population. Subjects with unsuccessful implant solely due to a failure to establish i2i communication at end of implant procedure will be included and imputed as failures. Subjects with unsuccessful implants due to reasons other than AV synchrony (e.g., cardiac anatomy) will be excluded from this analysis.

Template 



### Statistical Analysis Plan



#### 2.3.4 Secondary Safety Endpoint Analysis

The secondary safety endpoint evaluates the 3-month Aveir atrial LP related complication free rate (CFR<sub>A</sub>) based on the CEC adjudication of adverse events. The secondary safety endpoint will be tested if all the primary endpoints are met.

An atrial LP complication is defined as an atrial device- or procedure-related SADE. Complications that are exclusively related to the ventricular LP or its delivery/retrieval will not be considered atrial LP complications and will be excluded from this evaluation. Complications that cannot be exclusively determined to be related to the ventricular or atrial LP will be considered atrial LP complications (e.g. femoral access complications, embolism, etc.).

The secondary safety endpoint hypothesis is:

 $H_0$ : CFR<sub>A</sub>  $\leq 84\%$  vs.  $H_1$ : CFR<sub>A</sub> > 84%

where 84% is the performance goal.

The CFR<sub>A</sub> at 3 months will be estimated as a binomial proportion and one-sided 97.5% LCB of CFR<sub>A</sub> will be calculated using the normal approximation. The null hypothesis is rejected at the 2.5% significance level if the LCB exceeds the Performance Goal (PG) of 84%. The p-value from a one-sided Z-test for the binomial proportion will also be calculated and compared to the 0.025 significance level.

The primary analysis population for the secondary safety endpoint analysis will be based on subjects in the full analysis population, and the analysis will be conducted on all subjects with data available for the evaluation. Subjects who withdraw from the study or die prior to the 3-month follow-up visit (lower window) without an atrial complication will be excluded from this analysis. Atrial complications that occur through 3 months (90 days) will be included in the secondary safety endpoint analysis.

To eliminate the possible impact of Covid-19 on the secondary safety endpoint analysis, CEC adjudicated atrial complications that are related or possibly related to Covid-19 will be excluded. Additional analysis with these events included will also be provided.

#### 2.3.5 Secondary Effectiveness Endpoint Analysis

The secondary effectiveness endpoint includes evaluation of CAEP exercise protocol for atrial LP. The secondary effectiveness endpoint will be tested if all the primary endpoints are met, and the secondary Safety endpoint is also met.

The secondary effectiveness CAEP endpoint hypothesis is:

H<sub>0</sub>: Mean Slope < 0.65 or Mean Slope > 1.35

Template 



## Statistical Analysis Plan

 $H_1$ :  $0.65 \le Mean Slope \le 1.35$ .

#### CAEP exercise protocol

To demonstrate an appropriate and proportional response of sensor-indicated rate in graded exercise tests, all capable subjects who have completed the 6-minute walk test (6MWT) will be asked to perform a maximal effort CAEP exercise protocol. The subject will undergo the CAEP exercise test any time after the beginning of their 3-month visit window and before the end of 6-month visit window. Each subject will undergo this test at a single visit.

Data from subjects who have completed the 6MWT and have completed at least stage 3 of the CAEP exercise protocol, or 3.6 metabolic equivalent of task (METs), will be included in the analysis. Any CAEP assessments performed which substantially deviate from the CAEP exercise protocol or where insufficient data is available will be excluded from the analysis. The results of subjects who did not meet the analysis criteria will still be reported.

A mixed effects model for repeated measures will be used to estimate the mean slope (through origin) and standard error of mean slope across N subjects. A no intercept model with unstructured covariance matrix for the random effect (subject) will be used for this analysis. A 95% confidence interval for the mean slope will be provided and if this interval falls within the equivalence bounds of [0.65,1.35], the null hypothesis is rejected.



emplate 



## Statistical Analysis Plan



Up to thirty subjects will provide data contributing to this analysis. Based on recently reported studies of marketed rate-responsive pacemakers the expected slope for similar devices, including the Aveir device, is estimated to be approximately 77%, with an associated standard deviation of 14%. It is estimated based on these data that a sample size of 8 subjects would be sufficient to demonstrate that the lower and upper 95% confidence bounds meet the success criterion, based on a normally distributed random variable. To ensure that a robust cross-section of subjects is evaluated, however, a total of 30 subjects will undergo this assessment.

### 2.4 Sample Size Calculations



Template 



## Statistical Analysis Plan

| Powe | <u>ower calculation for the primary effectiveness endpoint #</u> | |
|---|---|---|
| | | able subjects wil |
| • | | 82.5% and reject the null hypothesis at a |
| 2.5% | 5% one-sided significance level. T | |
| Dowe | ower calculation for the primary effectiveness endpoint #2 | at 3 months (Rate) |
| 1 000 | 267 evaluab | |
| provid | | 83% and reject the null hypothesis at a 2.5% |
| • | ne-sided significance level. | |
| _ | | |
| Powe | ower calculation for the secondary safety endpoint at 3 m | |
| | | evaluable subjects performance goal of 84% and reject the null |
| hypot | /pothesis at a 2.5% one-sided significance level. T | performance goal of 64 % and reject the num |
| , | | |
| Additi | dditional sample size for the study | |
| | | up to 200 additional de |
| | ovo subjects will be enrolled<br>ssess the upgradeability to a Aveir DR LP system in subje | . Up to 50 subjects will also be enrolled t |
| | ngle chamber analysis. | icts previously implanted with the Aveil VK Li |
| omigic | ngie chamber analysis. | |
| 0.5 | | |
| 2.5 | 5 Interim Analysis | |
| 2.6 | 6 Timing of Analysis | |
| 0 = | | |
| 2.7 | 7 Study/Trial Success | |

emplate 



## Statistical Analysis Plan

### 2.8 Subgroups for Analysis

Subgroup analysis will be conducted for the primary safety and effectiveness endpoints (in the full analysis population) to assess consistency by gender on the following data:

-Gender: Male and Female

The data will be summarized, and 95% confidence interval will be reported for each gender group. The comparisons between the subgroups are not powered for hypothesis testing and are exploratory in nature.

Other subgroup analyses by age (< median and >=median) and select comorbidities with sufficient representation will also be performed using the same method as the subgroup analysis by gender.

## 2.9 Handling of Missing Data

A subject may discontinue from the study prior to the 3-month visit. If this situation occurs, reasons for missing data will be summarized to assess the plausibility if the missing data could affect subject's endpoint results.

In addition, sensitivity analyses will be performed to evaluate the potential impact of missing data on the primary safety and effectiveness endpoints.

#### Sensitivity Analyses for Primary Safety Endpoint

For the primary safety endpoint, tipping point analyses will be conducted on all the subjects in the full analysis population.

For the tipping point analysis,

#### Sensitivity Analyses for Primary Effectiveness Endpoint #1

The following sensitivity analysis will be conducted for the primary effectiveness endpoint #1.

Complete Case: Complete case sensitivity analysis will be conducted for subjects in the full analysis population

Tipping Point: Tipping Point sensitivity analysis will be conducted for subjects in the full analysis population.

Template 



## Statistical Analysis Plan

Sensitivity Analyses for Primary Effectiveness Endpoint #2

For the primary effectiveness endpoint #2, tipping point sensitivity analyses will be conducted in the full analysis population

### 2.10 Poolability Issue

Poolability of the primary safety endpoint and the two primary effectiveness endpoints on subjects in the full analysis population will be evaluated by region and across sites. Analysis will be performed based on available data.

The study will be conducted in up to 85 sites in the United States, Canada, Europe and Asia Pacific. The study will be conducted following the same investigational plan, monitoring plan and training plan in all regions. The consistency of results for the primary safety and effectiveness endpoints will be evaluated across regions i.e., US and OUS (outside the US) if there is a sufficient sample size in each region, and across sites with the following site categories:

Large sites: # of subjects enrolled ≥10 Medium sites: 4≤ # of subjects enrolled ≤9 Small sites: # of subjects enrolled ≤3

Descriptive summaries for the primary safety and the two primary effectiveness endpoints will be presented across (1) Regions: US or OUS (outside the US) and (2) Site Categories (Large, Medium or Small). Consistency of results will be examined using Fisher's exact test and assessed at a significance level of 0.15.

## 2.11 Multiplicity Issues

## 2.12 Adjustments for Covariates

l emplate 



## **Statistical Analysis Plan**

### 3.0 <u>DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA</u>

#### 3.1 Baseline and Demographic Characteristics

The following baseline, demographic, medical history and medication variables will be summarized descriptively for the subjects in the full analysis population: gender, age, ethnicity, race, history of smoking; key cardiovascular history, prior cardiac interventions, arrhythmia history, primary indication for study device implant, use of beta blocker, ACE, ARB, anti-coagulation, anti-arrhythmic, and anti-platelet medications, etc. and as needed. For subjects enrolled from European sites, race and ethnicity are not collected and hence will not be included in race/ethnicity summary of the demographics table.

#### 3.2 Adverse Events

All reported adverse events (AE), serious adverse events (SAE), adverse device effects (ADE), serious adverse device effects (SADE), unanticipated adverse device effect (UADE) or unanticipated serious adverse device effect (USADE) will be summarized for subjects in full analysis population using the number of events, the number of subjects with events and the percentage of subjects with events.

All CEC adjudicated events will also be summarized for subjects in full analysis population with the number of events, the number of subjects with events and the percentage of subjects with events. An AE listing which includes all adverse events and whether or not each event is device-related or procedure-related will be provided.

### 3.3 Subject Early Termination

Subject early termination reasons including deaths, withdrawals, lost-to-follow-up, etc. will be summarized at all scheduled visits.

#### 3.4 Protocol Deviation

Protocol deviations will be summarized by major and minor categories for subjects in whom a protocol deviation was reported.

#### 3.5 Additional Data

The following additional data will be recorded and reported descriptively:

- Comparisons of demographics between the study population to the existing dual-chamber pacemaker population by region using publicly available data
- All adverse events, and whether or not each is device-related or procedure-related
- Implant success rate and reasons for unsuccessful implant
- Device handling characteristics at implant
- Number of device repositioning at time of implantation
- Implant duration, fluoroscopy duration, and time from implant to hospital discharge
- Pre-procedure (i.e., MRI, CT, X-ray) and procedural imaging (i.e., ICE) measures to evaluate the right atrium and/or the atrial LP based on any imaging data provided to the Sponsor
- Final location of LP placement
- Demographics: gender, age, ethnicity, race, indication for pacemaker implant

Medical history

Template 



## Statistical Analysis Plan

- Use of beta blocker, ACE, ARB, anti-coagulation, anti-arrhythmic, and anti-platelet medications
- Remaining device longevity at the six-month visit, as displayed by the programmer based on delivered therapy, programmed settings, percent pacing, and measured pacing impedance.
- Average base rate, impedance, pulse amplitude, pulse duration and percentage pacing will also be reported for all visits
- Hospitalizations
- Mortality
- AV synchrony (at various positions and activity levels)
- Upgradeability of the Aveir ventricular LP (VR) into the Aveir DR LP system summarized by:
  - Success rate of VR to DR upgrades and reasons for unsuccessful upgrades.
  - Summary of adverse events related to upgrades
  - o Summary of device measurements for subjects with an upgrade
- EQ-5D Health-Related Quality of Life Analysis

#### 3.6 **24-Hour Holter Monitor Data Analysis**

All capable *de novo* subjects will be asked to wear a 24-hour Holter monitor and complete a symptom diary, until 50 subjects provide data contributing to the analysis. The test may be performed any time after the beginning of the 3-month visit window. The preferred window to perform the 24- hour Holter test is between the 3-month and 6-month visit. These data will be examined for appropriate sensing, pacing, AV Synchrony during the activities of daily living for each subject. In addition, these data will be evaluated for any correlation between any subject symptoms with losses of AV synchrony, if present.

A 24-hour Holter summary report will be provided which includes the following for each subject:

- Minimum, maximum, and average heart rate
- Percent atrial pacing
- A telemetry strip of the minimum heart rate and a telemetry strip during pacing (the pacing strip may be the same as the minimum heart rate strip but is not required).
- Number of pauses seen (defined as RR interval greater than or equal to 2 sec or < 30 bpm)
- All telemetry strips of a pause greater than the programmed lower rate limit after accounting for any hysteresis programming
- All telemetry strips showing evidence of atrial oversensing, undersensing, or loss of capture
- Programmed parameters (which are necessary to assess if the pauses or minimum heart rate seen on Holter are appropriate or not)
- AV Synchrony
- Appropriate Automatic Mode Switching (AMS) due to atrial arrhythmias
  Reported adverse events and/or subject symptoms with diary entry that is timed and dated to
  correlate Holter findings with events and/or symptoms.

Template 



## **Statistical Analysis Plan**

## 4.0 **DOCUMENTATION AND OHER CONSIDERATIONS**

All analyses will be performed using SAS® for Windows, version 9.2 or higher.

## 5.0 ACRONYMS AND ABBREVIATIONS

| Acronym or Abbreviation | Complete Phrase or Definition |
|---|---|
| CEC | Clinical Events Committee |
| IRB | Independent or institutional review board |
| EC | Ethics Committee |
| CIP | Clinical Investigation Plan |
| CRF | Case Report Form |
| AE | Adverse Event (Non-Serious Adverse Event) |
| SAE | Serious Adverse Event |
| ADE | Adverse Device Effect (Non-Serious Adverse Device Effect) |
| SADE | Serious Adverse Device Effect |
| UADE | Unanticipated Adverse Device Effect |
| USADE | Unanticipated Serious Adverse Device Effect |
| ACE | angiotensin-converting enzyme |
| ARB | angiotensin II receptor blocker |
| CFR | Complication-free rate |
| 6MWT | Six-minute walk test |
| CAEP | Chronotropic Assessment Exercise Protocol |
| MET | Metabolic Equivalent of Task |
| LCB | Lower Confidence Bound |
| AV | Atrioventricular |
| SAS | Statistical Analysis System |
| SAP | Statistical Analysis Plan |

## 6.0 **REFERENCES**

- ABT-CIP-10416/ Rev C, the CIP for Aveir DR i2i study
- CRD\_1023 Aveir DR Case Report Form

Template 



## Statistical Analysis Plan



Template 



## Statistical Analysis Plan

Template 



## Statistical Analysis Plan



Template



## **Statistical Analysis Plan**



Template 



## **Statistical Analysis Plan**



Template